CLINICAL TRIAL: NCT07180524
Title: Prospective Clinical Trial on the Impact of Uterine Fibromatosis Surgery on Pelvic Floor.
Brief Title: Prospective Clinical Trial on the Impact of Uterine Firomatosis on Pelvic Floor.
Status: Recruiting | Type: Observational
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Arsenio Spinillo, Principal Investigator, Fondazione IRCCS Policlinico San Matteo di Pavia
Other Study IDs: FIBROPELV
Record Dates: First submitted 2025-03-04; First posted 2025-09-18 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Pelvic Floor Dysfunction; Fibromatosis
MeSH Terms: conditions — Fibroma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- uterine fibromatosis: patinets with uterine fibromatosis will undergo hystrectomy or myomectomy

SUMMARY:
Uterine fibromatosis is one of the most frequent gynecological conditions; in fact, uterine fibroids involve approximately 25-30% of women during the fertile period. Risk factors for the development of this pathology include age, family history and ethnicity. Multiparity, advanced age for pregnancy and smoking appear to be protective factors.

Myomas are responsible for numerous symptoms reported by patients, such as menometrorrhagia, pelvic pain and urinary and/or deficatory symptoms. Although myomas are asymptomatic in almost 50% of cases, they represent the first cause of hysterectomy for benign pathologies (about 2/3 of cases). Urinary symptoms associated with myomas are rarely studied in patients with symptomatic uterine fibromatosis; therefore the impact that this pathology has on the symptoms related to pelvic-perineal dysfunction and what their prevalence is is not well known at present. The prevalence of urinary symptoms in women with uterine myomas is highly variable based on literature data and the studies considered; in fact, the most frequently reported urinary symptoms are urinary urgency (31-59%), dysuria (4-36%) and stress urinary incontinence (20-80%). Furthermore, there is currently no unanimous agreement between the topography and size of myomas and related urinary and pelvic symptoms.

The type of treatment varies from single or multiple myomectomy to hysterectomy performed laparoscopically or laparotomy. The choice of surgical approach depends on the number, size and position of myomas. To date, few studies have evaluated the impact of the type of surgical treatment on pelvic floor symptoms. In fact, although hysterectomy is considered a risk factor for the onset of pelvic floor disorders, removal of the uterus can sometimes improve urinary symptoms. However, some authors report, equally, a significant improvement in urinary symptoms after myomectomy. Further studies are needed to clarify the impact of myoma treatment on urinary symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic uterine fibromatosis with intramural and/or subserosal myomas identified by ultrasound and topographically mapped
* Patients with scheduled hysterectomy or myomectomy

Exclusion Criteria:

* suspicion of malignant lesion.
* active tumors
* previous history of chemotherapy or radiotherapy
* pregnancy
* age <18 years or >55 years (postmenopause)
* history of pelvic static disorders prior to surgery

Ages: 35 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients with symptomatic uterine fibromatosis and candidates for surgical treatment aged between 40 and 55 years will be consecutively enrolled.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-06-30 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
pelvic floor biometry | at baseline, immediately after the surgery, 1 month after surgery, 6 and 12 months after surgery
  Compare the pelvic floor well-being of patients undergoing total hysterectomy compared to those undergoing myomectomy at 1 month, 6 and 12 months after surgery.

SECONDARY OUTCOMES:
pelvic floor biometry | at baseline, immediately after the surgery, 1 month, 6 and 12 months after surgery
  Compare pelvic hiatus area, anteroposterior diameter, and transverse diameter over time in patients who underwent total hysterectomy compared to those who underwent myomectomy.
pelvic floor biometry | at baseline, immediately after the surgery, 1 month, 6 and 12 months after surgery
  Compare of the pelvic hiatus over time in patients who underwent total hysterectomy compared to those who underwent myomectomy.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Policlinico San Matteo, SC Ostetricia e Ginecologia 1, Pavia, Pavia, Italy

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Background] Shaffer RK, Dobberfuhl AD, Vu KN, Fast AM, Dababou S, Marrocchio C, Lum DA, Hovsepian DM, Ghanouni P, Chen B. Are fibroid and bony pelvis characteristics associated with urinary and pelvic symptom severity? Am J Obstet Gynecol. 2019 May;220(5):471.e1-471.e11. doi: 10.1016/j.ajog.2019.01.230. Epub 2019 Jan 31. PMID 30711512
- [Background] Dagur G, Suh Y, Warren K, Singh N, Fitzgerald J, Khan SA. Urological complications of uterine leiomyoma: a review of literature. Int Urol Nephrol. 2016 Jun;48(6):941-8. doi: 10.1007/s11255-016-1248-5. Epub 2016 Feb 27. PMID 26922066